CLINICAL TRIAL: NCT05874817
Title: Retrospective Assessment of Adverse Events-Related Healthcare Resource Utilization and Costs of Immune Checkpoint Inhibitor and Targeted Therapy for Adjuvant Treatment of Melanoma
Brief Title: Retrospective Assessment of AE-Related Healthcare Resource Utilization and Costs of Immune Checkpoint Inhibitor and Targeted Therapy for Adjuvant Treatment of Melanoma
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CTMT212AUS62
Record Dates: First submitted 2023-05-12; First posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
This was a retrospective cohort study using Truven Health Analytics' MarketScan Commercial Claims and Encounters and Medicare Supplement and Coordination of Benefit administrative claims databases. The analysis was conducted using the most recent 5 years of data from the database, 01 January 2015, to 28 February 2021 (study period). Included patients were followed for outcome evaluation from the index date (first prescription of treatment, immunotherapy [IO] or targeted therapy [TT] following diagnosis of non-metastatic malignant melanoma and evidence of first lymph node resection), until the first occurrence of end of continuous eligibility or end of the study period.

ELIGIBILITY:
Inclusion Criteria:

* Patients with at least one diagnosis of malignant melanoma of skin (The International Classification of Diseases, 9th Revision, Clinical Modification [ICD-9] codes: 172.0-172.9 or V10.82; ICD-10 (10th revision) codes: C43.0 C43.10, C43.11, C43.111, C43.112, C43.12, C43.121, C43.122, C43.20, C43.21, C43.22, C43.30 C43.31 C43.39 C43.4, C43.51, C43.52, C43.59 C43.60, C43.61, C43.62, C43.70, C43.71, C43.72, C43.8 C43.9 D03.0 D03.10 D03.11, D03.111, D03.112, D03.12, D03.121, D03.122, D03.20 D03.21 D03.22 D03.30 D03.39 D03.4 D03.51 D03.52 D03.59 D03.60 D03.61 D03.62 D03.70 D03.71 D03.72 D03.8 D03.9 Z85.820) anytime from the start of data collection until the start of study period.
* Patients with a procedure of first lymph node dissection or nodal basin ultrasound surveillance, per the National Comprehensive Cancer Network (NCCN) guidelines version 2.2020. The first lymph node dissection / nodal basin ultrasound surveillance signified that the patient was eligible to receive systemic treatment as adjuvant therapy.
* The first lymph node dissection or nodal basin ultrasound surveillance (index adjuvant date) must have had a diagnosis of malignant melanoma of skin within 6 months, to ensure that the dissection was related to melanoma.
* Patients with at least pharmacy or medical claim for the study drugs within 1 year on and after index date. The index date was the date of first prescription of study drug, IO (i.e., nivolumab, ipilimumab + nivolumab, pembrolizumab) or dabrafenib + trametinib.
* At least 18 years of age at the time of adjuvant treatment initiation.
* Patients with at least 6 months of continuous enrollment prior to the index date.
* Patients with at least 6 months of continuous enrollment after the index date.

Exclusion Criteria:

* Patients with a diagnosis of non-melanoma primary malignancy (ICD-9: 140.xx-165.xx, 170.xx-171.xx, 173.xx-195.xx, 200.xx-208.xx; ICD-10: C00.x - C14.x, C41.x, C49.x, C50, C51) during the 6 months pre-index period.
* Patients with chemotherapy or interferon alpha before index date.
* Patients with pregnancy (ICD-9: 630.xx-679.xx, V22.xx-V24.xx, V27.xx-V28.xx; ICD-10: O00 - O99) any time during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study
Sampling Method: Non-Probability Sample
Enrollment: 17517 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with adverse events (AEs) following first systemic adjuvant therapy | Up to 5 years

SECONDARY OUTCOMES:
Percentage of patients with AEs following first systemic adjuvant therapy completion/discontinuation | Up to 5 years
Healthcare resource utilization (HCRU) associated with AEs following first systemic adjuvant therapy | 30 days
Healthcare costs associated with AEs following first systemic adjuvant therapy | 30 days
HCRU associated with AEs following first systemic adjuvant therapy completion/discontinuation | 30 days
Healthcare costs associated with AEs following first systemic adjuvant therapy completion/discontinuation | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, East Hanover, New Jersey, United States